CLINICAL TRIAL: NCT01501539
Title: Prevention of Hypergranulation Tissue After Gastrostomy Tube Placement: A Randomized Controlled Trial of Hydrocolloid Dressings
Brief Title: Prevention of Hypergranulation Tissue After Gastrostomy Tube Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Katherine Barsness, MD, Attending Physician, Department of Surgery, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB # 2011-14460
Record Dates: First submitted 2011-12-20; First posted 2011-12-29 (Estimated); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Soft Tissue Inflammation
Keywords: Hypergranulation tissue; Gastrostomy tube; Hydrocolloid dressing; Silver hydrocolloid dressing; Gastrostomy tube dislodgement; Wound infection; Peristomal skin breakdown
MeSH Terms: conditions — Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard postop gastrostomy tube care (No Intervention): At the completion of the operative procedure for gastrostomy tube placement, the surgical incisions and the gastrostomy tube will be covered with dermabond, steristrips, and/or tegaderm dressings, according to surgeon preference. Standard postop gastrostomy tube care. Insertion site cleaned with soap and water. No dressing added.
- Standard hydrocolloid dressing (Experimental): At the completion of the operative procedure for gastrostomy tube placement, the surgical incisions will be covered with dermabond, steristrips, and/or tegaderm dressings, according to the surgeons preference. The gastrostomy tube will have a thin layer of hydrocolloid dressing (HD) placed around the gastrostomy tube. The HD will be changed once every other day fo the first 30 days after gastrostomy tube placement. After 30 days, care will revert to standard care.
  Interventions: Procedure: Standard Hydrocolloid Dressing
- Silver hydrocolloid dressing (Experimental): At the completion of the operative procedure for gastrostomy tube placement, the surgical incisions will be covered with dermabond, steristrips, and/or tegaderm dressings, according to surgeon preference. The gastrostomy tube will have a thin layer of silver hydrocolloid dressing (HD) placed around the gastrostomy tube. The silver HD will be changed once every other day for the first 30 days after gastrostomy tube placement. After 30 days, care will revert to standard care.
  Interventions: Procedure: Silver Hydrocolloid Dressing

INTERVENTIONS:
Procedure: Standard Hydrocolloid Dressing — Treatment placed over insertion site.
  Other Names: FDA Class II-K medical products; Hollister Wound Care (Hollister Incorporated)
  Arms: Standard hydrocolloid dressing
Procedure: Silver Hydrocolloid Dressing — Place dressing against skin under gastrostomy tube
  Other Names: FDA Class II-K medical products; Hollister Wound Care (Hollister Incorporated)
  Arms: Silver hydrocolloid dressing

SUMMARY:
The primary objective of this study is to compare the incidence of postoperative hypergranulation tissue formation after gastrostomy tube placement among children randomized to one of three treatments, in addition to measuring tube dislodgements and rates of resource utilization for complications.

DETAILED DESCRIPTION:
Hypergranulation tissue is one of the major immediate complications of gastronomy tube placement. This study aims to determine if using a foam dressing upon placement will prevent its formation, as it has been demonstrated as an effective treatment in healing hypergranulation tissue formation post-operatively. Study participants will be randomized into one of three treatments after gastronomy tube placement (1) standard care, (2) plain foam treatment or (3) silver foam dressing. These treatments will be applied for 30 days post-operatively in addition to standard care of cleaning the gastronomy site daily with soap and water, if assigned to foam intervention. All study materials are free for duration of 30 day intervention and participation will not interfere with routine post-operative care of gastronomy tube site. The total duration of trial will be 6 months and will not require additional study visits outside of routine care. The rate of G-tube dislodgements and associated outcomes will also be measured during the trial.

ELIGIBILITY:
Inclusion Criteria:

* Children between 1 month and 17 years of age who undergo gastrostomy tube placement by a member of the pediatric surgery faculty at Children's Memorial Hospital will be eligible for inclusion in this study.

Exclusion Criteria:

* Children undergoing gastrostomy tube placement by gastroenterology or interventional radiology at Children's Memorial Hospital.
* Mother or caregiver of the patient is currently pregnant, breastfeeding and/or planning on getting pregnant within the next 60 days (silver HD has not been studied in pregnant or breastfeeding women)

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 171 (Actual)
Dates: Start 2010-12; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
The primary outcome is to measure change in Hypergranulation tissue formation around Gastrostomy tube. | 2 time points: 2 weeks and 6 months post insertion.

SECONDARY OUTCOMES:
The secondary outcome is to measure change in visual assessment of postoperative condition of gastrostomy tube insertion site. | 2 timepoints: 2 weeks and 6 months post insertion.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine A Barsness, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Children's Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No